CLINICAL TRIAL: NCT03061487
Title: The Influence of Statin Treatment on Aneurysmatic Disease
Brief Title: Influence of Statins in Artery Aneurysms
Acronym: INSTANT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2016.04
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Statin; Aneurysm; Extracellular Matrix Alteration
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Patients affected by central and peripheral aneurismatic disease with maximum statin daily dose ( Atorvastatin 80 mg, Simvastatin 40 mg, Rosuvastatin 40 mg).
  Patients will undergo Open Surgical Treatment of Aneurysm (Aneurysmectomy).
  The investigation consist in:
  * taking a preoperative blood sample to evaluate the MMPs circulating levels
  * taking an aneurismatic vassel wall istological sample with an intraoperative biopsy to evaluate the tissue MMPs and miRNAs levels
  Interventions: Procedure: Open Surgical Treatment of Aneurysm (Aneurysmectomy)
- Group II: Patients affected by central and peripheral aneurismatic disease with minimum statin daily dose.
  Patients will undergo Open Surgical Treatment of Aneurysm (Aneurysmectomy).
  The investigation consist in:
  * taking a preoperative blood sample to evaluate the MMPs circulating levels
  * taking an aneurismatic vassel wall istological sample with an intraoperative biopsy to evaluate the tissue MMPs and miRNAs levels
  Interventions: Procedure: Open Surgical Treatment of Aneurysm (Aneurysmectomy)

INTERVENTIONS:
Procedure: Open Surgical Treatment of Aneurysm (Aneurysmectomy) — Aneurysmectomy is a surgical procedure in which a localized, dilated, weakened section of an artery (aneurysm) is removed (resected). The artery is either replaced with a synthetic graft, as seen in an aneurysm in the chest (thoracic aneurysm), abdomen (abdominal aneurysm) or leg (femoral or popliteal aneurysm).

SUMMARY:
The altered balance between the proteinases and their tissue inhibitors (TIMPS) is one of the pathogenetical mechanism of the aneurysmatic connective tissue degeneration. The increasement of protease, collagenase and elastase activity results indeed in a dramatic drop of collagen and elastin tissue and serum levels.Matrix Metalloproteinases (MMPs) are a group of proteolytic enzymes that along with their specific and non-specific inhibitors modulate the extracellular matrix composition. Recent studies have suggested an interesting role of microRNAs (miRNAs) in the regulation mechanisms of inflammation.

The aim of our study is to analyse the influence of statin treatment on aneurysmatic disease by monitoring MMPs and miRNAs in aneurysmatic wall tissue and MMps blood levels.

DETAILED DESCRIPTION:
The altered balance between the proteinases and their tissue inhibitors (TIMPS) is one of the pathogenetical mechanism of the aneurysmal connective tissue degeneration. The increase of protease, collagenase and elastase activity results indeed in a dramatic drop of collagen and elastin tissue and serum levels.

Vessels wall strength decrease is associated with the blood flow shear stress and affects negatively the walls integrity, causing the aneurysmatic vessel degeneration.

Matrix Metalloproteinases (MMPs) are a group of proteolytic enzymes that along with their specific and non-specific inhibitors modulate the extracellular matrix composition.

So far, 25 MMPs have been discovered, in particular, the ones that will be considered in this study are: MMP-2, MMP-9, and neutrophil gelatinase-associated lipocalin (NGAL) a related protein which is able to control MMP-9 activities.

Inflammation plays a central role in the pathogenetical pathway of aneurysmatic developement. Recent studies have suggested an interesting role of miRNAs in the regulation mechanisms of inflammation. miRNAs are short ribonucleic acid molecules usually composed of 20 to 25 nucleotides that can regulate mRNA transcription and protein translation by targeting the 3'-untranslated regions (3'-UTR) of target genes. miRNAs are involved in various physiological responses and pathological processes. Increasing evidence suggest that miRNAs are involved in inflammatory responses. In particular the ones that will be focused on this study are: miR-29b, miR-21, miR-181a, miR-150.

Very often, patients with aneurysmatic disease are under statin treatment. Some Statins (Atorvastatin, Simvastatin or Rosuvastatin) with pleiotropic effects may also play a protective role by conditioning the progression of the aneurysmatic degeneration.

The aim of our study is to analyse the influence of statin treatment on aneurysmatic disease by monitoring some MMPs and related molecules (MMP-2, MMP-9 and NGAL), miRNAs (the evaluation will be performed in aneurysmatic wall tissues and circulating blood levels).

Patients affected by central and peripheral aneurysmatic disease will be recruited and then divided in two groups based on the dosage of the statin treatment: the first group with maximum statin daily dose (Atorvastatin 80 mg, Simvastatin 40 mg, Rosuvastatin 40 mg), the second group with minimum statin daily dose. The latter will be defined as the control group.

Only patients which will fullfill the criteria to undergo surgical treatment will be recruited in the study in order to collect biological specimen of the aneurysmatic tissues .

The investigation consist in:

* taking a preoperative blood sample to evaluate the MMPs circulating levels
* taking an aneurysmatic vessel wall histological sample with an intraoperative biopsy to evaluate the tissue MMPs and miRNAs levels.

Previously, several studies suggested a role of MMPs (MMP-2 and MMP-9) and miRNAs in regulation of aneurysm developement, in particular miR29b, miR-181a, miR-21, miR-150.

The comparison between MMPs Levels in the study group and in the control group might highlight a role for MMPs level as a marker of aneurysmatic disease progression, consequently allowing the patient's stratification by analysing the risk of aneurysmatic evolution and growth.

ELIGIBILITY:
Inclusion Criteria:

* Patients under statins treatment with pleiotropic effect: Simvastatin, Rosuvastatin, Atorvastatin
* Patients underwent open aneurysm repair
* Age >18
* signing informed consent

Exclusion Criteria:

* Patients with chronic diseases such as liver diseases
* Pazient whith malignant diseases
* Recreational drug intake and alcohol abuse
* Intake of statins other than those under study or in combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by central and peripheral aneurysmal disease are going to be recruited and then divided in two groups based on the dosage of the statin treatment: the first group with maximum statin daily dose ( Atorvastatin 80 mg, Simvastatin 40 mg, Rosuvastatin 40 mg), the second group with minimum statin daily dose. The latter will be defined as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-02-26 (Estimated); Study Completion 2018-04-27 (Estimated)

PRIMARY OUTCOMES:
Evaluation of MMP-2, MMP-9 and NGAL levels in blood and aneurysms tissue | 1 year
  MMP-2, MMP-9 and NGAL will be studied in both groups. Elisa Testing will be used to analyze the blood samples and Western blot analysis will be used for the tissue samples.
Evalutation of miRNAs levels in blood and aneurysms tissue | 1 year
  Evaluation of miRNAs levels (in particular miR29b, miR-181a, miR-21, miR-150) will be studied in both groups. Stem-loop reverse-transcription PCR (RT-qPCR) method will be used for measuring individual microRNAs (miRNAs) in tissue and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano de Franciscis, M.D., Study Chair — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra R, Grande R, Montemurro R, Butrico L, Calio FG, Mastrangelo D, Scarcello E, Gallelli L, Buffone G, de Franciscis S. The role of matrix metalloproteinases and neutrophil gelatinase-associated lipocalin in central and peripheral arterial aneurysms. Surgery. 2015 Jan;157(1):155-62. doi: 10.1016/j.surg.2014.06.008. Epub 2014 Nov 1. PMID 25444221
- [Background] de Franciscis S, Mastroroberto P, Gallelli L, Buffone G, Montemurro R, Serra R. Increased plasma levels of metalloproteinase-9 and neutrophil gelatinase-associated lipocalin in a rare case of multiple artery aneurysm. Ann Vasc Surg. 2013 Nov;27(8):1185.e5-7. doi: 10.1016/j.avsg.2013.01.011. Epub 2013 Aug 26. PMID 23988549
- [Background] Serra R, Volpentesta G, Gallelli L, Grande R, Buffone G, Lavano A, de Franciscis S. Metalloproteinase-9 and neutrophil gelatinase-associated lipocalin plasma and tissue levels evaluation in middle cerebral artery aneurysms. Br J Neurosurg. 2014 May 5. doi: 10.3109/02688697.2014.913777. Online ahead of print. PMID 24799278
- [Background] Piechota-Polanczyk A, Demyanets S, Mittlboeck M, Hofmann M, Domenig CM, Neumayer C, Wojta J, Klinger M, Nanobachvili J, Huk I. The Influence of Simvastatin on NGAL, Matrix Metalloproteinases and Their Tissue Inhibitors in Human Intraluminal Thrombus and Abdominal Aortic Aneurysm Tissue. Eur J Vasc Endovasc Surg. 2015 May;49(5):549-55. doi: 10.1016/j.ejvs.2015.02.011. Epub 2015 Mar 21. PMID 25800096
- [Background] Maegdefessel L, Azuma J, Toh R, Merk DR, Deng A, Chin JT, Raaz U, Schoelmerich AM, Raiesdana A, Leeper NJ, McConnell MV, Dalman RL, Spin JM, Tsao PS. Inhibition of microRNA-29b reduces murine abdominal aortic aneurysm development. J Clin Invest. 2012 Feb;122(2):497-506. doi: 10.1172/JCI61598. Epub 2012 Jan 24. PMID 22269326
- [Background] Adam M, Raaz U, Spin JM, Tsao PS. MicroRNAs in Abdominal Aortic Aneurysm. Curr Vasc Pharmacol. 2015;13(3):280-90. doi: 10.2174/15701611113119990015. PMID 23713862